CLINICAL TRIAL: NCT05433636
Title: Idle Waiting or Meditating: Does a Brief, Mindfulness Intervention in the Clinic Waiting Room Improve Patient Outcomes?
Brief Title: Mindful Waiting Room
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00085446_AM_00042941
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Anxiety State; Depressive State; Pain; Nausea; Fatigue; Cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain; Nausea; Fatigue; Neoplasms | interventions — Whole Body Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Body Scan Practice (Experimental)
  Interventions: Behavioral: Body Scan
- Mindful Breathing Practice (Experimental)
  Interventions: Behavioral: Mindful Breathing
- Mindfulness of Discomfort Practice (Experimental)
  Interventions: Behavioral: Mindfulness of Discomfort
- Mindful Savoring Practice (Experimental)
  Interventions: Behavioral: Mindful Savoring
- Integrative Health Recording (Active Comparator)
  Interventions: Behavioral: Integrative Health Recording

INTERVENTIONS:
Behavioral: Body Scan — Patients will listen to a 5-minute, audio-recorded body scan practice.
  Arms: Body Scan Practice
Behavioral: Mindful Breathing — Patients will listen to a 5-minute, audio-recorded mindful breathing practice.
  Arms: Mindful Breathing Practice
Behavioral: Mindfulness of Discomfort — Patients will listen to a 5-minute, audio-recorded mindfulness of discomfort practice.
  Arms: Mindfulness of Discomfort Practice
Behavioral: Mindful Savoring — Patients will listen to a 5-minute, audio-recorded mindful savoring practice.
  Arms: Mindful Savoring Practice
Behavioral: Integrative Health Recording — Patients will listen to a 5-minute, audio-recorded description of integrative health.
  Arms: Integrative Health Recording

SUMMARY:
This will be a single-site, five-arm, parallel group randomized control trial involving patients seeking integrative healthcare. Four different styles of 5-minute, audio-recoded mindfulness practices delivered in the clinic waiting room will be compared with a 5-minute audio-recording about integrative healthcare.

A secondary sub-analysis will investigate the most effective mindfulness practice style for patients presenting at the clinic with elevated anxiety, depression, or pain.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment at the Huntsman Cancer Institute's Wellness Center
* Adults 18+
* Facility with the English language that is adequate to complete study procedures

Exclusion Criteria:

* Cognitive impairment preventing completion of study procedures
* An unstable illness judged by medical staff to interfere with study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-09-14 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | A single 5-minute period
  75% of patients that begin an audio recording will listen to the full, 5-minute recording

SECONDARY OUTCOMES:
Change in Pain | Immediately before to after 5-minute audio recording
  Single item assessing pain ("Right now, I feel physical pain") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater pain.
Change in Anxiety | Immediately before to after 5-minute audio recording
  Single item assessing anxiety ("Right now, I feel nervous, anxious or on edge") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater anxiety.
Change in Depression | Immediately before to after 5-minute audio recording
  Single item assessing depression ("Right now, I feel down, depressed, of uninterested in life") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater depression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States